CLINICAL TRIAL: NCT06683365
Title: A Phase I Study of the Feasibility and Safety of SuraL nervE Tissue Grafting to the Substantia nigrA in Patients With Synucleinopathies (LEAP)
Brief Title: Autologous suraL nervE Grafting to the Substantia nigrA in Patients With Synuclienopathies
Acronym: LEAP
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Craig van Horne, MD, PhD (Other)
Collaborators: University of Kentucky CCTS (Unknown)
Responsible Party: Sponsor-Investigator, Craig van Horne, MD, PhD, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 95534; UL1TR001998 (NIH)
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Multiple System Atrophy; Parkinsons Disease
Keywords: Synucleinopathies; Cell and Tissue Based Therapy; Multiple System Atrophy; Parkinsons Disease
MeSH Terms: conditions — Multiple System Atrophy; Parkinson Disease; Synucleinopathies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nerve Graft Recipients (Experimental)
  Interventions: Procedure: Sural Nerve Graft to the Substantia Nigra
- Placebo Group (Placebo Comparator)
  Interventions: Procedure: Sham surgery

INTERVENTIONS:
Procedure: Sural Nerve Graft to the Substantia Nigra — Participants assigned to this arm will have the sural nerve biopsied from one of their ankles. This cellular tissue will be deposited bilaterally into the substantia nigra area of their brain by a specialized cannula via bilateral scalp incisions and skull burr holes.
  Arms: Nerve Graft Recipients
Procedure: Sham surgery — Participants assigned to this arm will have the sural nerve from one of their ankles biopsied in the same fashion as the experimental arm. Bilateral incisions will be made on the participants scalp but no burr holes into the skull and no cannula passes into the brain will occur.
  Arms: Placebo Group

SUMMARY:
This phase I double-blind study focuses on the safety and feasibility of implanting autologous peripheral nerve tissue (PNT) into the substantia nigra area of the brain in persons who have been diagnosed with either Parkinson's disease (PD) or Multiple System Atrophy (MSA). 7 participants will be enrolled, with 4 participants receiving the graft and 3 receiving a sham surgery. Eligible participants will be early in their diagnosis with a lower burden of symptoms. Participants will be followed initially for one year after surgery.

DETAILED DESCRIPTION:
This phase I double blind clinical trial will be used to plan future, larger clinical trials that would test how autologous cells from the peripheral nerve may help in the repair of damaged brain cells in Parkinson's Disease (PD) or Multiple System Atrophy (MSA) and slow the progression of the diseases. We will be judging the feasibility of implanting a participant's own cells from a nerve in the leg into the substantia nigra area of the brain. Patients eligible for participation will be at an earlier in stage of the disease with symptoms being less severe and therefore would not yet qualify for DBS. The LEAP trial is a study where the first participant will receive an implantation of the cells from their own sural nerve (a nerve near the ankle), into the substantia nigra on both sides of their brain. The 6 participants who follow, will be randomized to one of two arms. The 3 participants assigned to the experimental arm will receive the graft. The 3 participants assigned to the control arm will receive a sham surgical procedure, where the sural nerve will be biopsied, and bilateral scalp incisions will be made. Those who do not receive the cells initially may be eligible to undergo another surgery at the end of the study, after un-blinding has occurred, to receive the cell implants.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of clinically established or clinically probable PD or MSA as defined by MDS criteria
* Disease duration greater than 2 years
* Age 40-75, inclusive
* MDS-Unified Parkinson's Disease Rating Scale (UPDRS) Part III greater than or equal to 20 points but less than or equal to 35 points, off anti-parkinsonian medication for PD or MDS-Unified Multiple System Atrophy Rating Scale (UMSARS) less than or equal to 30 points off anti-parkinsonian medication
* No MDS-UPDRS Part III score >3 on items 3.3, 3.4, 3.5, 3.6, 3.7, 3.8, 3.14 while off medication
* Able and willing to undergo ioflupane/SPECT
* Able to tolerate the surgical procedure
* Able to undergo all planned assessments
* Available access to the sural nerve

Exclusion Criteria:

* Previous PD surgery or intracranial surgery
* Ongoing major medical or psychiatric disorder incl. depression and psychosis
* Other concomitant treatment with neuroleptics
* Typical, nonparkinsonian syndrome ioflupane/SPECT signal
* Unable to undergo an MRI
* An obstructed trajectory path to the substantia nigra
* Significant microvascular disease
* Use of anticoagulants other than aspirin
* Female who is pregnant, lactating, or of child-bearing potential unwilling to use an adequate birth control method during the period of the study
* Consent capacity will be assessed and determined during and throughout a participant's neuropsychological exam. A participant who experiences a decline in consent capacity prior to surgery, will be removed from the study by the PI. A decline in consent capacity after surgery will not result in the removal of the participant in the study.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2028-12-02 (Estimated); Study Completion 2030-12-02 (Estimated)

PRIMARY OUTCOMES:
Meet recruitment goal | Trial opening through 12 months
  Ability to recruit, enroll, and assign participants to the trial within 12 months of the trial opening.

SECONDARY OUTCOMES:
Study-related serious adverse events as assessed by MedDRA v.27 | Enrollment through 12 months
  Total number of serious adverse events associated with bilateral PNT collection and deployment to the substantia nigra. Serious adverse events will be defined as an abscess, tumor, infection of the bed of the graft, altered mental state, seizure, ankle or foot infection, wound dehiscence at the ankle incision, spread of neuropathy of the ankle or foot on the ipsilateral side of the nerve biopsy, or other event determined by the PI/investigators to be important.
Study-related adverse events as assessed by MedDRA v27 | Enrollment through 6 month study visit
  Total number of adverse events experienced by participants categorized by System Organ Class and/or High Level Group Term using MedDRA v27 for designation.
Number of deployment attempts required to deliver bilateral PNT | During the procedure
  Per protocol, the surgeon has two chances to successfully deploy 60% of the PNT tissue loaded in the guide-tube into the brain per hemisphere. The number of attempted deployments will be documented and if <60% of the tissue is deployed after two attempts, a failed delivery will be documented and no other attempts will be made.
Duration of procedure | During the procedure
  Number of minutes it takes for the procedure to be completed. This will be defined by the anesthesia start time and anesthesia end time.
Length of hospital admission | Admission for the procedure through hospital discharge
  The number of days each participant is admitted to the inpatient hospital for the procedure and acute post-operative care.
Percent of study visit completed by participants | Enrollement through 12 month study visit
  The number of designated study visits completed compared to the total number of study visits that are scheduled to occur.
Change in Neuropsychological diagnosis | Baseline and 12 months
  Changes in participant neuropsychological diagnoses during scheduled evaluations will be reported. e.g. No cognitive diagnosis progressing to mild neurocognitive disorder.
Mean change in Neuropsychological assessment scores | Baseline to 12 months
  Participants complete a neuropsychological assessment battery that meets the MDS guidelines for determining mild cognitive impairment/mild neurocognitive disorder. Domains include attention and working memory, executive functioning, memory (verbal and visual), language, and visuospatial skills. Participants' raw scores will be converted to standardized scores based on appropriate norms (e.g., age-based norms). Participants' 12 month re-evaluation will be compared to their baseline pre-surgical assessment to determine change from baseline on each measure. A change that exceeds 1.5 standard deviation from their baseline performance will be considered notable.
Mean change in Montreal Cognitive Assessment (MoCA) scores | Baseline, 4 weeks, 6 months, and 12 months
  Mean change in MoCA scores for participants at study visits compared to baseline by group allocation. Assessment is scored from 0-30 with a score of 26 or better indicating normal cognition. A score less than 26 indicates a cognitive deficit.
Mean change of the Movement Disorder Society - Unified Parkinsons Disease Rating Scale (MDS-UPDRS) Part I scores | 4 weeks, 6 and 12 months as compared to baseline
  MDS-UPDRS Part I scores non-motor symptoms effecting activities of daily living in those with Parkinson's Disease. Scores range from 0-52 with higher scores indicating greater symptom severity.
Mean change of the MDS-UPDRS Part II scores | 4 weeks, 6 months, and 12 months compared to baseline
  MDS-UPDRS Part II scores motor symptoms effecting activities of daily living in those with Parkinson's Disease. Scores range from 0-52 with higher scores indicating greater symptom severity.
Mean change in MDS-UPDRS Part III scores | 4 weeks, 6 and 12 months compared to baseline
  MDS-UPDRS Part III scores motor symptoms associated with Parkinson's Disease. Part III scores range from 0-132 with higher scores indicating higher symptom severity.
Mean change in MDS-UPDRS Part IV scores | 4 weeks, 6 and 12 months compared to baseline
  MDS-UPDRS Part IV scores motor complications such as fluctuations and dyskinesia's associated with anti-Parkinson's medications. Scores range from 0-24 with higher scores indicating greater severity in motor complications.
Mean change of the Movement Disorder Society - Unified Multiple System Atrophy Rating Scale (MDS-UMSARS) Part I scores | 4 weeks, 6 and 12 months as compared to baseline
  MDS-UMSARS Part I rates patient reported functional disabilities. Scores for this section range from 0-48 with higher scores indicating greater disability
Mean change of the MDS-UMSARS Part II scores | 4 weeks, 6 months, and 12 months compared to baseline
  MDS-UMSARS Part II scores motor symptoms associated with multiple system atrophy. Scores range from 0-56 with higher scores indicating greater symptom severity.
Mean change in MDS-UMSARS Part III scores | 4 weeks, 6 and 12 months compared to baseline
  MDS-UMSARS Part III assesses orthostatic hypertension symptoms. This part examines blood pressure changes when a participant stands up after laying down for two minutes. It is scored as either a "Yes" the participant experiences orthostatic hypertension, or a "No" the participant does not don't experience orthostatic hypertension.
Mean change in MDS-UMSARS Part IV scores | 4 weeks, 6 and 12 months compared to baseline
  MDS-UMSARS Part IV assess the participants global disability. Scores range from 1-5 with 1 being completely independent and 5 being totally dependent/bedridden.
Mean change in Parkinson's Disease Questionnaire-8 (PDQ-8) quality of life scores | Monthly through 12 month study visit compared to baseline
  Assess changes in participant's quality of life. Questionnaire is scored from 0-32 with higher scores indicating poorer quality of life.
Mean change in Modified Schwab and England Scale of Activities of Daily Living scores | At 6 and 12 months compared to baseline
  Mean change participant independence levels as measured in Schwab and England Scale of Activities of Daily Living scores. 100% = completed independent and 0% being completely dependent.
Mean change in Non-motor symptom scale scores | Baseline and 12 months
  Assessment used to identify Parkinson's disease related non-motor symptoms experienced by participants. The scale measures the frequency and severity of symptoms and is scored from 0-360 with higher scores indicating more frequent and severe symptoms.
Participants electing to receive Deep Brain Stimulator (DBS) | Enrollment through 12 month study visit
  Number of study participants who elect to have DBS implanted prior to completing the 12 month study visit.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
Images and results may be made available to other researchers by asking participants, at the time of consent, their willingness to permit sharing of data and bio-specimens.

REFERENCES:
- [Result] Quintero JE, Slevin JT, Gurwell JA, McLouth CJ, El Khouli R, Chau MJ, Guduru Z, Gerhardt GA, van Horne CG. Direct delivery of an investigational cell therapy in patients with Parkinson's disease: an interim analysis of feasibility and safety of an open-label study using DBS-Plus clinical trial design. BMJ Neurol Open. 2022 Jul 14;4(2):e000301. doi: 10.1136/bmjno-2022-000301. eCollection 2022. PMID 35949912
- [Result] van Horne CG, Quintero JE, Gurwell JA, Wagner RP, Slevin JT, Gerhardt GA. Implantation of autologous peripheral nerve grafts into the substantia nigra of subjects with idiopathic Parkinson's disease treated with bilateral STN DBS: a report of safety and feasibility. J Neurosurg. 2017 Apr;126(4):1140-1147. doi: 10.3171/2016.2.JNS151988. Epub 2016 May 6. PMID 27153166
- [Result] van Horne CG, Quintero JE, Slevin JT, Anderson-Mooney A, Gurwell JA, Welleford AS, Lamm JR, Wagner RP, Gerhardt GA. Peripheral nerve grafts implanted into the substantia nigra in patients with Parkinson's disease during deep brain stimulation surgery: 1-year follow-up study of safety, feasibility, and clinical outcome. J Neurosurg. 2018 Dec 1;129(6):1550-1561. doi: 10.3171/2017.8.JNS163222. Epub 2018 Feb 18. PMID 29451447